CLINICAL TRIAL: NCT02627040
Title: A Prospective Randomized Trial of Intertrochanteric Femoral Fractures Treated With a Single Screw Versus a Two-integrated Screw Cephalo-medullary Nail.
Brief Title: Intertrochanteric Femoral Fracture Fixation Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Florida Orthopaedic Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00023144
Record Dates: First submitted 2015-11-25; First posted 2015-12-10 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Intertrochanteric Fracture; Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- InterTan Intertrochanteric Nail (Active Comparator): 'Surgical fixation' of intertrochanteric fracture with a cephalomedullary nail with an InterTan device (two-integrated screws)
  Interventions: Device: InterTan Intertrochanteric Nail
- Gamma 3 Intertrochanteric Nail (Active Comparator): 'Surgical fixation' of intertrochanteric fracture with a cephalomedullary nail and Gamma 3 locking nail (single screw)
  Interventions: Device: Gamma 3 Intertrochanteric Nail

INTERVENTIONS:
Device: InterTan Intertrochanteric Nail — Cephalomedullary fixation of intertrochanteric fracture with an InterTan Intertrochanteric Nail
  Arms: InterTan Intertrochanteric Nail
Device: Gamma 3 Intertrochanteric Nail — Cephalomedullary fixation of intertrochanteric fracture with an Gamma 3 Intertrochanteric Nail
  Arms: Gamma 3 Intertrochanteric Nail

SUMMARY:
The main goal of the study is to determine which cephalomedullary nail results in a better functional outcome for the patient with an unstable intertrochanteric hip fracture. Subjects will be randomized to fixation with either a Gamma3 cephalomedullary nail or an InterTan cephalomedullary nail. Outcomes will be reviewed over a 12 month follow-up period.

DETAILED DESCRIPTION:
Primary Hypotheses:

Patients who maintain their initial fracture reduction and subsequent position over time with minimal femoral neck shortening and varus will demonstrate significantly improved functional abilities, including gait and abductor function.

Secondary Objective:

* Whether radiographic differences in femoral neck shortening and varus collapse translate into a worse functional outcome to the patient.
* Whether there are differences in mortality between treatments
* Whether there is a time frame follow up after which there is no difference in outcomes.
* Evaluate the device used for fracture stabilization as a potentially contributing factor for maintenance of normal or near-normal abductor function and gait.

Primary Outcome:

The primary outcome will be functional abilities at 3, 6 and 12 months after injury. The following measures of functional ability will be utilized:

Methods:

This is a prospective, randomized non-blinded study. Patients will be identified as they present to the orthopaedic trauma service of Tampa General Hospital with a qualifying injury to determine their interest in participating in the study. Written informed consent will be obtained prior to initiation of any study procedures.

Group A will undergo cephalomedullary nail-based single screw intertrochanteric hip fracture fixation device (Gamma 3 nail). Group B will receive the integrated dual screw intertrochanteric hip fracture fixation device (Intertan nail). Patient outcomes will be analyzed using intention to treat principles. Following randomization assignment, surgeons will all follow the identical described surgical technique, with the only variable being the implant used. Post-operative immobilization and time to weight bearing and rehabilitation protocols will be again identical for all patients regardless of fixation technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients surgically treated for an intertrochanteric femur fracture at Tampa General Hospital.

  * Skeletally mature patients over the age of 60; both genders.
  * Community ambulators.

Exclusion Criteria:

* Patients with ipsilateral lower extremity injury
* Patients under age 60
* Co-existent, severe knee or back problems
* Muscle contracture around the knee or hip joint
* Individuals who have had TKA within 6 months
* Body mass index (BMI; kg/m2) >40
* Suspicious of pathologic fracture (tumor in origin)
* Pre-op mobility: Non ambulatory; ambulatory indoors with living support
* Cognitive impairment or dementia
* Prisoners or impending incarceration
* Homeless or no stable address.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2015-11-30 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Hip Function | 6 months post-operatively
  Hip Function measured with Harris Hip Score.

SECONDARY OUTCOMES:
Functional outcome | 6 months post-operatively
  Functional outcome will be measured using the following outcome measurement: Gait analysis using MiniSun's IDEEA® LifeGait System, a portable device for assessment of functional gait outcomes.
Walking ability | 3 months post-operatively
  Subjects will wear a pedometer applied in the immediate post-operative period, and will continue to wear it for 3 months. Total walking steps will be measured.
Hip range of motion | 6 months post-operatively
  Range of motion of hip measured with Harris Hip Score.
Hip Pain | 6 months post-operatively
  Pain measured with Harris Hip Score.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan R Mir, MD, MBA, Principal Investigator — Florida Orthopaedic Institute
Locations (2):
- United States (2):
  - Brandon Regional Hospital, Brandon, Florida
  - Tampa General Hospital, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data.